CLINICAL TRIAL: NCT02389322
Title: Phase IIb Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 on Healthy People Aged 18-65,Adopting Randomized Blinded and Parallel Controlled Method
Brief Title: Phase IIb Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 on Healthy People Aged 18-65
Acronym: IIb-healthy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Air Force Military Medical University, China (Other); Proswell Medical Corporation (Industry); Jiangsu Province Centers for Disease Control and Prevention (Network); Jurong Province Centers for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EC-IIb-healthy
Record Dates: First submitted 2015-03-05; First posted 2015-03-17 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2015-09

CONDITIONS: Tuberculosis
Keywords: ESAT6; CFP10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5μg/ml ESAT6-CFP10 after BCG immunization (Experimental): A within group paired comparison of 5μg/ mL ESAT6-CFP10 and TB-PPD in 48 person of study population II. The 5μg/ mL ESAT6-CFP10 and TB-PPD agents are given concomitantly to each volunteer in the right and left forearms 12 weeks after BCG immunization, according to a randomisation scheme .
  Interventions: Biological: 5μg/ml ESAT6-CFP10; Biological: BCG
- 10μg/ml ESAT6-CFP10 after BCG immunization (Experimental): A within group paired comparison of 10μg/ mL ESAT6-CFP10 and TB-PPD in 48 person of study population II. The 10μg/ mL ESAT6-CFP10 and TB-PPD agents are given concomitantly to each volunteer in the right and left forearms 12 weeks after BCG immunization, according to a randomisation scheme .
  Interventions: Biological: 10μg/ml ESAT6-CFP10; Biological: BCG
- 5μg/ml ESAT6-CFP10 after placebo immunization (Placebo Comparator): A within group paired comparison of 5μg/ mL ESAT6-CFP10 and TB-PPD in 48 person of study population II. The 5μg/ mL ESAT6-CFP10 and TB-PPD agents are given concomitantly to each volunteer in the right and left forearms 12 weeks after placebo controlled immunization, according to a randomisation scheme .
  Interventions: Biological: placebo
- 10μg/ml ESAT6-CFP10 after placebo immunization (Placebo Comparator): A within group paired comparison of 10μg/ mL ESAT6-CFP10 and TB-PPD in 48 person of study population II. The 10μg/ mL ESAT6-CFP10 and TB-PPD agents are given concomitantly to each volunteer in the right and left forearms 12 weeks after placebo controlled immunization, according to a randomisation scheme.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: 5μg/ml ESAT6-CFP10 — The participants are injection intradermally with 0.1 ml 5μg/ml ESAT6-CFP10 12 weeks after BCG immunization or placebo immunization.This biological diagnostic reagents is injection agent .Every subject apply for the 5μg/mlRecombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 only one time after choosing into study population II .
  Other Names: 5μg/mlEC
  Arms: 5μg/ml ESAT6-CFP10 after BCG immunization
Biological: 10μg/ml ESAT6-CFP10 — The participants are injection intradermally with 0.1 ml 10μg/ml ESAT6-CFP10 12 weeks after BCG immunization or placebo immunization.This biological diagnostic reagents is injection agent .Every subject apply for the 10μg/mlRecombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 only one time after choosing into study population II .
  Other Names: 10μg/ml EC
  Arms: 10μg/ml ESAT6-CFP10 after BCG immunization
Biological: BCG — The participants are injected intradermally with 0.1 ml BCG.This BCG is Freeze-dried agent and with five people dose of each bottle,so each bottle of BCG must dissolve by 0.5ml special diluent before administration.Every subject apply for the BCG vaccine only one time after choosing into study population II .
  Other Names: Bacillus Calmette-Guerin
  Arms: 10μg/ml ESAT6-CFP10 after BCG immunization; 5μg/ml ESAT6-CFP10 after BCG immunization
Biological: placebo — The participants are injected intradermally with 0.1 ml placebo of Bacillus Calmette-Guerin.This placebo is Freeze-dried agent and with five people dose of each bottle ,so each bottle must dissolve by 0.5ml special diluent before administration.Every subject apply for the BCG vaccine only one time after choosing into study population II .
  Arms: 10μg/ml ESAT6-CFP10 after placebo immunization; 5μg/ml ESAT6-CFP10 after placebo immunization

SUMMARY:
The investigators select 500 subjects who meet the standard and are considered as study population I. Do specific gamma-interferon detection before the skin test， then inject intradermally with two dosage ESAT6-CFP10 and Tuberculin purified protein derivative (TB-PPD) at different arm of the same subject and get 192 participants whose three kinds of detection result are all negative and are considered as study population II.Then,they are immune to the Bacillus Calmette-Guerin (BCG) vaccine or the placebo of the BCG. Do specific gamma-interferon detection before the skin test， then inject intradermally with two dosage ESAT6-CFP10 and TB-PPD at different arm of the same subject 12 weeks after immunity.Negative rate of ESAT6-CFP10 after vaccination BCG as the main index , evaluate the specificity of different doses of ESAT6-CFP10, and conform the optimal dose of ESAT6-CFP10.

DETAILED DESCRIPTION:
1.the correlation of three detection methods for study population I

500 study population I are randomly divided into two different dose group on average, according to ESAT6-CFP10 dose(5μg/ml or 10μg/ml). Do specific gamma-interferon(γ-IFN) detection before the skin test，then inject intradermally with 5μg/ml ESAT6-CFP10 or 10μg/ml ESAT6-CFP10 and TB-PPD at different arm of the same subject.Evaluate respectively the positive rate of three detection methods 、the correlation of three detection methods and the security of study population I after application for ESAT6-CFP10 .

2.screen study population II

Choose those participants, whose result of three detection (ESAT6-CFP10、TB-PPD andγ-IFN ) all negative, HIV negative and chest X-ray no abnormalities, into study population II.

3.study population II vaccinate BCG or placebo

Study population II ,according to the same proportion ,are randomly divided into four group in double blinded state,: 5μg/ml ESAT6-CFP10 after BCG immunization, 10μg/ml ESAT6-CFP10 after BCG immunization, 5μg/ml ESAT6-CFP10 after placebo-controlled immunization , 10μg/ml ESAT6-CFP10 after placebo-controlled immunization.They vaccinate BCG or the placebo of BCG.

4.Inject ESAT6-CFP10 12 weeks after inoculation in study population II

The investigators draw blood and operate specific gamma-interferon(γ-IFN) detection before the skin test，then inject intradermally with 5μg/ml ESAT6-CFP10 or 10μg/ml ESAT6-CFP10 (in double blinded state) and TB-PPD at different arm of the same subject ,according to the above grouping scheme.

Calculate the negative coincidence rate and the correlation of three detection methods, and observe the safety of ESAT6-CFP10 in study population II at the same time.Evaluate the specificity of different doses of ESAT6-CFP10, negative rate of ESAT6-CFP10 after vaccination BCG as the main index. And finally conform the optimal dose of ESAT6-CFP10.

ELIGIBILITY:
* Inclusion Criteria of study population Ⅰ:

  1. 18 to 65 years old;
  2. Consent and signed informed consent forms(ICF);
  3. Comply with follow-up;
  4. No history of tuberculosis;
  5. Physical condition : No obvious heart, liver, kidney, gastrointestinal tract, nervous system, mental disorder and metabolic abnormalities and other medical history from signed informed consent to the injection within four weeks prior to delivery ;by the comprehensive physical examination showed electrocardiogram, blood pressure, heart rate, breathing and laboratory tests, including blood, urine routine, liver, kidney and other various biochemical test all without exception or slightly unusual but does not affect our research;
  6. Normal axillary temperature(quiet condition ≤37.0 ℃).
* Inclusion Criteria of study population Ⅱ:

  1. healthy people conforming to the study population Ⅰ criteria ;
  2. the result of three detection methods( ESAT6-CFP10 (5 μg/ml or 10 μg/ml)、 TB - PPD and specific gamma - IFN ) are all the negative ;
  3. Comply with two criteria the above (1) (2) , HIV negative, X-ray chest radiograph no abnormalities.

Exclusion Criteria of study population Ⅰand study population Ⅱ:

1. Has the following serious disease, such as advanced cancer, diabetes, chronic obstructive pulmonary disease (copd) in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc;
2. Have epilepsy, brain and nervous system symptoms or signs of history or have risk tendency of epilepsy, brain and other nervous system disease and not easy to control;
3. Has known or suspected (or risk possible) immune damaged or abnormal functional , accept glucocorticoid and immunosuppressants or immunopotentiator treatment, outside the gastrointestinal tract protein or blood products or plasma extraction in 3 months, immunodeficiency virus infection or related diseases or long-term use of antibiotics;
4. Has acute febrile diseases and infectious diseases;
5. taking part in any other new drug clinical trials or participated in any other new drug clinical trials within 3 months before this trials;
6. allergy to drugs 、alcohol 、 vaccine、drugs using in this experiment and allergic or scar constitution;
7. In pregnancy or lactation;
8. With mental or physical disabilities;
9. Researchers consider that any conditions may affect the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
immune response of ESAT6-CFP10 from the size of induration or redness in all population | within 72 Hours After Intradermal Injection With ESAT6-CFP10
  We measure the size 24h,48h,72h after administered intradermally ESAT6-CFP10
immune response of TB-PPD from the size of induration or redness in all population | within 72 Hours After Intradermal Injection With TB-PPD
  We measure the size 24h,48h,72h after administered intradermally TB-PPD
the results of specificity γ-IFN test in all subjects | before administered intradermally

SECONDARY OUTCOMES:
the Number of Participants With Adverse Events | within 72 hours after injection
ESAT6-CFP10 cosistency with TB-PPD in all subjects | within 72 hours after injection
ESAT6-CFP10 cosistency with γ-IFN in all subjects | within 72 hours after injection
TB-PPD cosistency with γ-IFN in all subjects | within 72 hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, Master, Principal Investigator — Jingsu Province Centers for Disease Control and Prevention
Locations (1):
- Jurong Province Centers for Disease Control and Prevention, Jurong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- [Derived] Xu M, Lu W, Li T, Li J, Du W, Wu Q, Liu Q, Yuan B, Lu J, Ding X, Li F, Liu M, Chen B, Pu J, Zhang R, Xi X, Zhou R, Mei Z, Du R, Tao L, Martinez L, Lu S, Wang G, Zhu F. Sensitivity, Specificity, and Safety of a Novel ESAT6-CFP10 Skin Test for Tuberculosis Infection in China: 2 Randomized, Self-Controlled, Parallel-Group Phase 2b Trials. Clin Infect Dis. 2022 Mar 1;74(4):668-677. doi: 10.1093/cid/ciab472. PMID 34021314
- See also: Center for drug evaluation,China Food and Drug Administration(CFDA) ,China — https://wbca.cde.org.cn/wbca/clinmain.do?method=edit&ckmIdCode=8BE5738082A97A9E5471F80B4F814FCF